CLINICAL TRIAL: NCT05056311
Title: Engaging Families to Improve the Care of Patients With Hypospadias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Indiana University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-0146; K23DK111987 (NIH)
Record Dates: First submitted 2021-08-31; First posted 2021-09-24 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: Hypospadias
Keywords: hypospadias; shared decision making; decisional regret; decision aid
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent Utilization of Decision Aid Website (Experimental): All enrolled parents will view the decision aid website for as long and as frequently as they wish before the initial visit to the urologist.
  Interventions: Other: Decision Aid Website

INTERVENTIONS:
Other: Decision Aid Website — The (private) decision aid website contains information in text, graphic, and video form about hypospadias and considerations for choosing surgery and no surgery.

SUMMARY:
Reconstructive surgery is advocated for most children with hypospadias, a condition in which the pee hold is not in the correct place on the penis, to prevent potentially serious cosmetic and functional problems. Parents faced with a decision about hypospadias repair encounter an irreversible choice with potentially lifelong consequences. Recent studies have identified decisional conflict (DC) and decisional regret (DR) as a significant problem for parents. Several recent guidelines on complex urologic topics suggest that shared decision-making (SDM) is the optimal approach.

A pilot test of a decision aid website by parents potentially facing this decision will be conducted to measure pre- and post-outcomes, in order to develop a fuller understanding of how urologists can effectively provide parents with optimal decision support. Parents will answer questions via phone up to four time points, twice before (T1 and T2) and twice after seeing a urologist for a hypospadias referral (T3 and T4). If the urologist diagnoses hypospadias but recommends no surgery, the final data collection point will be three months after the urology visit. If the urologist recommends repair surgery, the final data collection point will be six months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* parents 18 years of age and older of sons with hypospadias, or a tentative hypospadias diagnosis, and/or referral to a urologist for hypospadias
* patient newborn up to age 5 years
* parent able to consent and do interview in English
* parent access to a reliable internet and smart phone, tablet, or computer to view the website
* child/patient scheduled to see a urologist, but must not have yet seen the urologist at the time of enrollment
* parent aware that there is an issue with child's pee hole
* parent planning to attend urology appointment

Exclusion Criteria:

* As target enrollment groups are filled, parents may be excluded in order to achieve a balanced sample, e.g. exclusion of mothers/female caregivers.

Ages: 0 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hubert Chan, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - UNC, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parent Utilization of Decision Aid Website
Started | 65
Received Intervention | 64
Completed | 27
Not Completed | 38
Not completed — Lost to Follow-up | 14
Not completed — Withdrawal by Subject | 1
Not completed — Dropped from study due to no Hypospadias | 23

BASELINE CHARACTERISTICS:
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 49
  More than one race | 2
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64
Child's Age at Consent [Mean (Standard Deviation); unit: days] | 149 (197)
Child's Meatal Location (Confirmed hypospadias) [Count of Participants; unit: Participants] — Population: Only 30 children were diagnosed with hypospadias at the consultation with the urologist.
  Participants
    number analyzed (Participants) | 30
    Glanular (includes megameatus) | 15
    Distal Shaft | 10
    Mid Shaft | 3
    Penoscrotal | 2
    Perineal | 0
Marital Status [Count of Participants; unit: Participants]
  Single | 26
  Married | 33
  Separated | 1
  Divorced | 3
  Widowed | 0
  Other | 1
Education [Count of Participants; unit: Participants]
  Some High School | 4
  Graduated High School | 13
  Some College | 19
  College Degree | 22
  Post-Graduate Degree | 6
Health Insurance [Count of Participants; unit: Participants]
  Public (Medicaid/Children's Special Services/TBC) | 28
  Private (Anthem/Aetna/TBC) | 19
  Other insurance type/unknown | 9
  Self-pay | 8
Health Literacy [Count of Participants; unit: Participants] — Participants were asked: "How often do you need to have someone help you when you read instruction, pamphlets, or other written material from your doctor or pharmacy?"
  Participants
    Never | 39
    Rarely | 13
    Sometimes | 8
    Often | 2
    Always | 2
Mean Income by Zip Code [Mean (Standard Deviation); unit: dollars annually] | 55900 (18000)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eligible Parents Screened (Feasibility)
Description: Recruitment is defined as the number of potential participants who are eligible divided by the total number screened multiplied by 100.
Time Frame: Baseline (T1)
Population: All available data are reported. Data reported for parents who were screened for eligibility.
Measure: Number; unit: percentage of parents recruited
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 148
percentage of parents recruited | 90.5

2. Primary Outcome: Percent of Eligible Parents Enrolled (Feasibility)
Description: The number of parents enrolled divided by the total number of parents who were eligible multiplied by 100.
Time Frame: Baseline (T1)
Population: All available data are reported. Data reported for eligible parents.
Measure: Number; unit: percentage of parents enrolled
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 134
percentage of parents enrolled | 48.5

3. Primary Outcome: Decision Aid Acceptability by Categories of Information, Length, Clarity, and Balance (Acceptability)
Description: Acceptability of a decision aid refers to ratings regarding the comprehensibility of components of a decision aid, its length, clarity, amount of information, and balance in presentation of information about options. The tool has 4 questions with answers on a Likert scale ranging from 1-5 (length, amount of information, and balance) and 1-4 (clarity). A response of 3 is ideal for information, length, and balance and a response of 1 is ideal for clarity.
Time Frame: Pre-consultation, 1 week after baseline (T2)
Population: All available data are reported. Between T1 and T2, 9 parents were lost to follow up and 1 parent withdrew from the study for a total of 54.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 54
Participants
  Information : Much less than wanted | 0
  Information : A little less than wanted | 4
  Information : About right | 38
  Information : A little more than wanted | 7
  Information : Much more than wanted | 5
  Length: Much too long | 1
  Length: A little too long | 2
  Length: About right | 45
  Length: A little too short | 5
  Length: Much too short | 1
  Clarity: Everything was clear | 16
  Clarity: Most things were clear | 34
  Clarity: Some things were clear | 3
  Clarity: Many things were unclear | 1
  Balance: Clearly slanted to surgery | 3
  Balance: Slightly slanted to surgery | 10
  Balance: Completely balanced | 38
  Balance: Slightly slanted to no surgery | 3
  Balance: Clearly slanted to no surgery | 0

4. Primary Outcome: Percentage of Parents Retained in the Study (Feasibility)
Description: Number of parents who completed the study divided by the number of eligible parents enrolled who completed the study multiplied by 100.
Time Frame: T1 to T4, a total of approximately 6 months
Population: All available data are reported. Of the 64 parents who completed T1, 9 were lost to follow up and 1 withdrew. Of the 54 who completed T2, 1 parent was lost to follow up before the consultation. Of the 53 completing the consultation, 23 were found to not to have hypospadias. Of the 30 patients diagnosed with hypospadias, 1 parent was lost to follow up prior to T3. Of the 29 parents who completed T3, 2 parents were lost to follow up prior to T4 resulting in a total of 27 parents who completed T4.
Measure: Number; unit: percentage of participants
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 64
percentage of participants | 42.2

5. Secondary Outcome: Mean Decisional Conflict Scale (DCS) Score at T1 and T2
Description: The Decisional Conflict Scale (DCS) measures personal perceptions of uncertainty in choosing options, modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making, and effective decision making (in full version) such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. This study utilizes the full version, a Likert-type scale consisting of 16 questions and answer options of strongly agree to strongly disagree. Total scores range from 0-100, a higher score means more decisional conflict.
Time Frame: Baseline (T1), Pre-consultation, 1 week after baseline (T2)
Population: All available data are reported. Data reported includes participants who completed the Decisional Conflict Scale for T1, T2, and T3. Between T1 and T2, 9 parents were lost to follow up and 1 parent withdrew from the study for a total of 54. Of the 54, 1 parent was lost to follow up prior to provider consultation. After completing the consultation, 23 were diagnosed without hypospadias and were discontinued.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 54
score on a scale
  T1 | 35.97 (18.81)
  T2: number analyzed (Participants) | 29
  T2 | 21.93 (11.84)
Statistical Analysis 1: Comparison: Parent Utilization of Decision Aid Website; Test type: Superiority; p = 0.001, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

6. Secondary Outcome: Mean Decisional Conflict Scale (DCS) Score at T2 and T3
Description: The Decisional Conflict Scale (DCS) measures personal perceptions of uncertainty in choosing options, modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making, and effective decision making (in full version) such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. This study utilizes the full version, a Likert-type scale consisting of 16 questions and answer options of strongly agree to strongly disagree. Total scores range from 0-100, a higher score means more decisional conflict. Time frame revised to address original entry error.
Time Frame: Pre-consultation, 1 week after baseline (T2), Initial post-consultation, within 48 hours of urology visit (T3)
Population: All available data are reported. Between T1 and T2, 9 parents were lost to follow up and 1 parent withdrew from the study for a total of 54. Of the 54, 1 parent was lost to follow up prior to provider consultation. Of the 53 who completed the consultation, 23 were found to not to have hypospadias and were discontinued. One parent was lost to follow up during T3, resulting in 29.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 29
score on a scale
  T2 | 21.93 (11.84)
  T3 | 8.78 (9.61)
Statistical Analysis 1: Comparison: Parent Utilization of Decision Aid Website; Test type: Superiority; p = 0.001, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

7. Secondary Outcome: Mean Decision-Specific Knowledge Scores
Description: Decision-Specific Knowledge is a six-question tool with multiple choice question and answer options created by the investigator to measure pre/post knowledge of hypospadias and repair surgery. Total scores range from 0-100% with a higher score indicating more correct answers.
Time Frame: Baseline (T1), Pre-consultation, 1 week after baseline (T2)
Population: All available data are reported. 64 participants completed the baseline decision-specific knowledge quiz but 10 did not complete the pre-clinic decision-specific knowledge quiz. Between T1 and T2, 9 parents were lost to follow up and 1 parent withdrew from the study. Scores are reported for 54 participants who completed the baseline and pre-clinic decision-specific knowledge quiz.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parent Utilization of Decision Aid Website: All enrolled parents will view the decision aid website for as long and as frequently as they wish before the initial visit to the urologist. Decision Aid Website: The (private) decision aid website contains information in text, graphic, and video form about hypospadias and considerations for choosing surgery and no surgery.
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 54
score on a scale
  T1 | 54.32 (22.24)
  T2 | 75.62 (16.42)
Statistical Analysis 1: Comparison: Parent Utilization of Decision Aid Website; Test type: Superiority; p = 0.001, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

8. Secondary Outcome: Mean Decisional Regret Scale Score
Description: The Decision Regret Scale measures distress or remorse after a decision. Brehaut's (2003) 5-item scale has scores ranging from 0-100, where 100 indicates maximal regret, and 0 indicates no regret.
Time Frame: 3-month post-consultation (T4)
Population: All available data are reported. Between T1 and T2, 9 parents were lost to follow up and 1 parent withdrew from the study for a total of 54. Of the 54, 1 parent was lost to follow up prior to provider consultation. After completing the consultation, 23 were diagnosed without hypospadias and were discontinued. One parent was lost to follow up during T3. Two parents were lost to follow up between T3 and T4 totaling 27.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 27
score on a scale | 25.0 (47.03)

9. Secondary Outcome: Hypospadias Treatment Preference by Category at T1 and T2
Description: This is a single question created by the investigator asking "Do you intend for your son to have hypospadias surgery?" with yes/no/unsure answer options to measure a change in response, or not, after viewing the decision aid website.
Time Frame: Baseline (T1), Pre-consultation, 1 week after baseline (T2)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 64
Participants
  T1: Yes | 31
  T1: No | 2
  T1: Unsure | 31
  T2: number analyzed (Participants) | 54
  T2: Yes | 27
  T2: No | 2
  T2: Unsure | 25
Statistical Analysis 1: Comparison: Parent Utilization of Decision Aid Website; Test type: Superiority; p = 0.0001, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

10. Secondary Outcome: Hypospadias Treatment Preference by Category at T2 and T3
Description: as for outcome 9
Time Frame: Pre-consultation, 1 week after baseline (T2), Initial post-consultation, within 48 hours of urology visit (T3)
Population: All available data are reported. Between T1 and T2, 9 parents were lost to follow up and 1 parent withdrew from the study for a total of 54. Of the 54, 1 parent was lost to follow up prior to provider consultation. After completing the consultation, 23 were diagnosed without hypospadias and were discontinued. One parent was lost to follow up during T3.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 54
Participants
  T2: Yes | 27
  T2: No | 25
  T2: Unsure | 2
  T3: number analyzed (Participants) | 29
  T3: Yes | 18
  T3: No | 1
  T3: Unsure | 10
Statistical Analysis 1: Comparison: Parent Utilization of Decision Aid Website; Test type: Superiority; p = 0.6374, McNemar — The a priori threshold for statistical significance was <0.05

11. Secondary Outcome: Awareness of Decision by Category at T1 and T2
Description: This is a single question created by the investigator asking "Is there a decision to make about whether your son should have surgery for his hypospadias?" with yes/no/unsure answer options to measure a change in awareness of decision, or not, after viewing the decision aid website.
Time Frame: Baseline (T1), Pre-consultation, 1 week after baseline (T2)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 64
Participants
  T1: Yes | 37
  T1: No | 6
  T1: Unsure | 21
  T2: number analyzed (Participants) | 54
  T2: Yes | 34
  T2: No | 0
  T2: Unsure | 20

12. Secondary Outcome: Awareness of Decision by Category at T2 and T3
Description: as for outcome 11
Time Frame: Pre-consultation, 1 week after baseline (T2), Initial post-consultation, within 48 hours of urology visit (T3)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 54
Participants
  T2: Yes | 34
  T2: No | 20
  T2: Unsure | 0
  T3: number analyzed (Participants) | 29
  T3: Yes | 20
  T3: No | 1
  T3: Unsure | 8

13. Secondary Outcome: Mean Shared Decision Making Questionnaire Score
Description: The Shared Decision Making Questionnaire measures the decisional process in medical encounters from both the patient and the physician perspectives. The questionnaire contains 9 questions with answers on a 6-point Likert scale. Scores range from 0-100 with higher scores indicating a higher perceived level of shared decision making.
Time Frame: Initial post-consultation, within 48 hours of urology visit (T3)
Population: All available data are reported. Between T1 and T2, 9 parents were lost to follow up and 1 parent withdrew from the study for a total of 54. Of the 54, 1 parent was lost to follow up prior to provider consultation. After completing the consultation, 23 were diagnosed without hypospadias and were discontinued. One parent was lost to follow up before T3, resulting in 29 parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 29
score on a scale | 82.5 (16.7)

14. Secondary Outcome: Mean Preparation for Decision Making Score
Description: The Preparation for Decision Making scale (Prep-DM) scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation focused on making a health decision. The scale contains 10 questions with answers on a Likert Scale Scores range from 0-100 with higher scores indicating a higher perceived level of preparation for decision making.
Time Frame: Pre-consultation, 1 week after baseline (T2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Utilization of Decision Aid Website
Number analyzed (Participants) | 54
score on a scale | 82.6 (14.1)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion. Enrollment occured from 1 week up to 6 months before the initial urology visit through. Study completion occurred approximately 3 months post urology visit if no surgery or 6 months post surgery.
Arm/Group | Parent Utilization of Decision Aid Website
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT05056311/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT05056311/ICF_001.pdf